CLINICAL TRIAL: NCT06893653
Title: COMBINED EFFECTS OF FOCAL MUSCLE VIBRATION AND tDCS ON MOTOR RECOVERY IN STROKE
Brief Title: Focal Muscle Vibration and tDCS on Motor Recovery in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MalihaREC02168
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: stroke; tDCS; motor activity; spasticity
MeSH Terms: conditions — Stroke; Motor Activity; Muscle Spasticity | interventions — Transcranial Direct Current Stimulation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FMV (Active Comparator): FMV + PT
  Interventions: Device: Focal muscle vibration; Other: Physical Therapy
- tDCS (Active Comparator): tDCS + PT
  Interventions: Device: tDCS; Other: Physical Therapy
- FMV & tDCS (Active Comparator): FMV + tDCS + PT
  Interventions: Other: Physical Therapy; Device: Focal muscle vibration & tDCS
- PT (Active Comparator): PT only
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Device: Focal muscle vibration — FMV will be applied to the muscle belly along with the conventional physical therapy
  Arms: FMV
Device: tDCS — tDCS will be applied to M1 area of brain along with the conventional physical therapy
  Arms: tDCS
Other: Physical Therapy — Conventional physical therapy will be provided
Device: Focal muscle vibration & tDCS — Focal muscle vibration with tDCS and conventional physical therapy will be provided.
  Arms: FMV & tDCS

SUMMARY:
Although tDCS and FV have shown some benefit as stand-alone treatment, researcher suggest that combining intervention with complementary mechanism can lead to additive or synergistic benefits which might yield more significant improvement in functional outcome hence the author propose to plan the combination of FV with tDCS for motor recovery /spasticity in stroke patients.

DETAILED DESCRIPTION:
A stroke is a medical condition characterized by a sudden, localized, loss of neurological function resulting from damage to the blood vessels in the central nervous system. It is a prevalent condition globally and leading cause of disability impairing motor function and significantly impact daily activities and work. 26% of individuals with stroke have a disability in ADLS and 50% have motor impairment gait disorder contribute to 20 to 30%. Spasticity 25%-40% which ultimately affect the quality of life of patients.

Spasticity arises from central nervous system damage where the loss of cortical neurons reduces descending inhibitory control over the spinal cord, affecting the balance between inhibitory and excitatory inputs leading to disinhibition of spinal reflexes causing hyperexcitability of stretch reflexes increase H reflex activity and impaired reciprocal inhibition.Fastest city interacts with weakness resulting in disabling motor impairments and complex complication like muscle contractor motor dysfunction and plastic paint which negatively impacts on patients quality of life.

Noninvasive brain stimulation (NIBS) has been seen more common in rehabilitation setting as an add on therapy to conventional rehabilitative treatment. The main goal of NIBS is to create neuromodulation by inhibiting or activating neural activity in the targeted cortical region. There are different modalities used for NIBS most widely used are transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS). tDCS involves a small current to the scalp aiming to modulate cortical excitability. Typical configuration of tDCS are the anode electrode place over the brain area of interest aiming to increase excitation and the cathode electrode placed as a reference, over contra lesional hemisphere aiming to decrease excitability and all electrode taste as a reference such as if she does not supra orbital region. In stroke recovery tDCS is often used to either enhance excitability in the lesioned hemisphere or suppress in the non-lesioned hemisphere to rebalance neural activity. The core concept of tDCS is operating on a simple principle, i.e. the positive terminal of the battery also referred to as the anode is connected to one special location on the head and the negative terminal or cathode is attached at the other end of the head. An electromotive force is generated between these two contact points on the head that creates a potential difference. This difference push positively charged ions that are potassium, sodium and calcium away from the anode towards the cathode this when way neurons that are located under the anode get a boost for excitation and at the same time inhibition occurs at the cathode and that's how whole brain activity is modulated.

Another intervention strategy that has potential for sustainable stroke rehabilitation is the use of mechanical vibration as a therapeutic intervention known as vibration therapy. Focal vibration (FV) reduces muscles spasticity, facilitate muscle contraction and stimulates the proper system to obtain efficient motor control during functional activities. In FV, mechanical vibrations are applied to localized muscles generally the muscle belly or the tendon on the affected side. The suggested mechanism of action of focal vibration on spasticity is depression of the H-reflex within the spinal motor neuron and reciprocal inhibition between the agonist and antagonist muscles.

A study was done aimed to assist the current evidence on the effect of tDCS on upper limb motor function and identified evidence suggest that tDCS has a superior effect in improving function of upper lamp in patient who had a stroke. In 2019, meta-analysis was done to explore the effect of tDCS on different stages of stroke (acute, sub-acute, chronic) and result show that tDCS had a significant effect in the patient of chronic group. Stronger connectivity of ipsilesional and the parietal cortex and contra lesional frontotemporal cortex was found to be associated with an increase in cortico spinal excitability following the anodal tDCS in chronic stroke survivors. A meta-analysis of multiple session reviewed how tDCS parameters influence upper limb function and demonstrate that tDCS applied during therapy yield significant results.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke
* Spasticity > 1 at Modified Ashworth Scale.
* FMA score more than 36

Exclusion Criteria:

* Metallic implant including shunt, intracranial pacemaker, surgical clip etc.
* Any neurological disorder other than stroke
* Any Orthopedic impairment that limit the motor recovery

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyr Assessment | 20th week
  FMA is used for the assessment of physical performance and sensorimotor function of neurological patients. It uses a 3-point ordinal scale to score individuals' ability to perform a certain task. Total score is 226. It has excellent inter and intrarater reliability
Modified Ashworth Scale | 20th week
  MAS is a tool to measure hypertonia. It scores the resistance on a 5 point ordinal scale with an increase value indicating hypertonia. Intrarater reliability of MAS was found to be good to excellent for upper (k= 0.71-0.94) and lower extremities(k= 0.55-0.97) while interrater reliability was poor to moderate for upper (k= 0.25-0.66) and lower extremities

SECONDARY OUTCOMES:
Stroke Specific Quality of Life questionnaire | 20th week
  It is used for estimating the quality of life of stroke patients. It contains 49 questions related to different personal and social aspects. Scoring is done on a ordinal scale of 1-5 with an increase score indicating independence. It is a valid and reliable tool to use in stroke population

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow AD, Shin J, Wang H, Kellawan JM, Pereira HM. Influence of Transcranial Direct Current Stimulation Dosage and Associated Therapy on Motor Recovery Post-stroke: A Systematic Review and Meta-Analysis. Front Aging Neurosci. 2022 Mar 18;14:821915. doi: 10.3389/fnagi.2022.821915. eCollection 2022. PMID 35370603
- [Background] Wang H, Yu H, Liu M, Xu G, Guo L, Wang C, Sun C. Effects of tDCS on brain functional network of patients after stroke. IEEE Access. 2020 Nov 13;8:205625-34
- [Background] Wang H, Chandrashekhar R, Rippetoe J, Ghazi M. Focal muscle vibration for stroke rehabilitation: a review of vibration parameters and protocols. Applied Sciences. 2020 Nov 21;10(22):8270